CLINICAL TRIAL: NCT04356417
Title: Long-term Use of Drugs That Could Prevent the Risk of Serious COVID-19 Infections or Make it Worse: Cases of Synthetic Antimalarial Drugs and Anti-hypertensive Drugs
Brief Title: Long-term Use of Drugs That Could Prevent the Risk of Serious COVID-19 Infections or Make it Worse
Acronym: TRAPSAH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GIS EPI-PHARE (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP200412
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: AMD, ACEi's/ARB Prevent/Worsen Risk of COVID-19 Infection
Keywords: Prevent COVID-19 infection; Synthetic antimalarial drugs (AMD); Anti-hypertensive drugs (ACEi's/ARB); SNSD; PMSI; Cohort
MeSH Terms: interventions — Angiotensin Receptor Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: - Synthetic anti-malarial drugs — Prevalent users will be those with at least one dispensing of AMD or ARBs/ACEi's from 01/01/2019 to 01/01/2020. Exposed users will be those among prevalent users who still received AMD or ARBs/ACEi's on 31/12/2019. The inclusion period will be from 01/01/2019 to 01/01/2020. The study end date will be 30/06/2020. For each treatment AMD or ARB/ACRi's, the persistence of treatment will be defined as the length of time from initiation to discontinuation. Initiation will be the date of the first reimbursement of AMD or ARB/ACRi's during the inclusion period. We will define the discontinuation of treatment as a period of more than 90 days without fulfilment of a prescription for the same treatment after the period covered by the previous prescription i.e 30 days. Exposure to a combination of drugs will be defined as a period shorter than 30 days between the prescription of two different systemic drugs and the fulfilment of another prescription for both drugs in the following 90 days.
  Other Names: - Converting enzyme inhibitors and angiotensin receptor antagonists

SUMMARY:
The COVID-19 emerging disease due to a novel coronavirus (SARS-CoV-2), started in Wuhan, China, last December, 2019. In the past three months, the virus has spread rapidly worldwide to reach the pandemic threshold.

Research has since been carried out and is intensifying in order to describe the clinical characteristics of infected patients, to identify the prognostic factors of acute respiratory distress syndrome [ARDS] and the death; and to assess the effectiveness of new antivirals and therapeutic strategies to treat COVID-19.

Treatments currently being investigated include:

* Potentially effective treatments: (hydroxy)chloroquine, Remdesivir, Lopinavir, Ritonavir +/- IFN-ß-1a (currently evaluated in the European discovery trial), methylprednisolone in patients with ARDS;
* Potentially harmful treatments: antihypertensives such as converting enzyme inhibitors and angiotensin receptor antagonists.

We made the hypothesis that (1) patients receiving ARBs or ACEi's have a higher risk to present a serious COVID-19 infection disease and (2) patients receiving synthetic AMD (e.g. HCQ and CQ) have a lower risk to present a serious covid19 infection disease.

Using data from the French insurance health database (SNDS) and hospital discharge database (PMSI), our objectives are

* Main objective: To assess the risk of moderate to serious COVID-19 infections in patients using synthetic anti-malarial drugs (AMD) or anti-hypertensive drugs (Angiotensin receptor-blocking/Angiotensin-converting-enzyme inhibitors).
* Secondary objective : To examine the risk of moderate to serious COVID-19 infections according of age, sex, co-morbidities, level of exposure of AMD, geographical locations and underlying comorbidities.

This in order to:

* To prevent moderate to serious COVID-19 infections in at-risk population (diabetes, elderly, respiratory failure population) using synthetic AMD.
* To prevent moderate to serious COVID-19 infections in at-risk population stopping angiotensin receptor-blocking and angiotensin-converting-enzyme inhibitors.

DETAILED DESCRIPTION:
Details for "Study design" section

Time perspective : Retrospective and prospective cohort study using French National Health Database Data source

Enrollment:

* 70,000 patients treated by synthetic AMD
* 13 million patients treated by ARBs or ACEi's from the French national health insurance database (SNDS) and the French national hospital discharge database (Programme de Médicalisation des Systèmes d'Information, PMSI)

ELIGIBILITY:
Inclusion Criteria:

All adults (18 years of age and older) registered in the French national health insurance database (SNDS) receiving between January 1, 2020, and May 31, 2020:

1. Synthetic anti-malarial drugs (AMD): Participants will be identified by the prescription of at least one synthetic AMD (chloroquine and hydroxychloroquine, ATC P01D1 and M01C respectively)
2. Anti-hypertensive drugs: Participants will be identified by the prescription of at least one Angiotensin receptor-blocking or Angiotensin converting- enzyme inhibitors, ATC C09A-D

No Exclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Refer to eligibility criteria
Sampling Method: Probability Sample
Enrollment: 6000000 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Identification of serious COVID-19 infections | From 2020/01/01 to 2020/06/30
  Participants as those with the emergency ICD-10 (international classification of diseases, 10th revision) code of U07.1 which was assigned to the disease diagnosis of COVID-19.

SECONDARY OUTCOMES:
Pneumonia infections | From 2020/01/01 to 2020/06/30
ICU stay | From 2020/01/01 to 2020/06/30
Oro-tracheal intubation | From 2020/01/01 to 2020/06/30
Death | From 2020/01/01 to 2020/06/30

CONTACTS AND LOCATIONS:
Overall Officials: Emilie SBIDIAN, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION